CLINICAL TRIAL: NCT00002148
Title: Parallel Group, Placebo-Controlled, Tolerability, Safety, and Efficacy Study of OPC-14117 in HIV Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 242A; 02-D94
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: Cognitive Disorders; HIV Infections
Keywords: Cognition Disorders; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Free Radical Scavengers; Antioxidants; OPC 14117
MeSH Terms: conditions — Cognitive Dysfunction; HIV Infections; Cognition Disorders; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — OPC 14117

INTERVENTIONS:
Drug: OPC 14117

SUMMARY:
To assess the tolerability and safety of OPC-14117. To evaluate effects of OPC-14117 on cognitive function, quality of life, and activities of daily living.

DETAILED DESCRIPTION:
Patients receive OPC-14117 or placebo bid for 12 weeks, followed by 12 weeks of open label therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity.
* Cognitive impairment.

Prior Medication:

Allowed:

* Prior OPC-14117 other than on the current study.
* Antiretroviral therapy if stable for 6 weeks prior to study entry (12 weeks for stavudine).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current opportunistic CNS infection (i.e., toxoplasmosis or cryptococcal meningitis).
* Severe pre-morbid psychiatric illness including schizophrenia and major depression that would interfere with protocol compliance.
* CNS neoplasms.
* Any other clinically significant condition or laboratory abnormality that would interfere with ability to participate on study.
* Current participation in other drug studies.

Patients with the following prior conditions are excluded:

* Past history of opportunistic CNS infection (i.e., toxoplasmosis or cryptococcal meningitis).
* History of chronic neurological disorders such as serious head injury, documented stroke, multiple sclerosis, uncontrolled epilepsy, Tourette's syndrome, and other neurodegenerative processes such as Huntington's disease.
* History of adverse reaction / allergy to OPC-14117.
* Prior participation on this study.

Prior Medication:

Excluded:

* Other investigational drugs within the past 30 days. Alcoholism within past 6 months (more than 2 drinks daily).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Columbia Univ, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York

REFERENCES:
- [Background] Safety and tolerability of the antioxidant OPC-14117 in HIV-associated cognitive impairment. The Dana Consortium on the Therapy of HIV Dementia and Related Cognitive Disorders. Neurology. 1997 Jul;49(1):142-6. doi: 10.1212/wnl.49.1.142. PMID 9222182